CLINICAL TRIAL: NCT01977235
Title: An Open, Randomized, Parallel Control, Multiple-center Phase II Trial of Two Different Dosages of Irinotecan Combined With Cisplatin Scheme in Extensive Disease-Small Cell Lung Cancer
Brief Title: Two Different Dosages of Irinotecan Combined With Cisplatin Scheme in Extensive Disease-Small Cell Lung Cancer
Acronym: TDICC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xueqin Yang, associate chief physician, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDICC
Record Dates: First submitted 2013-10-15; First posted 2013-11-06 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Irinotecan; Cisplatin; Small-cell lung cancer; UGT1A1
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Irinotecan 90mg/m2/iv over 90min and cisplatin 30mg/m2/iv over 60min on day 1 and 8, repeat Q 3weeks. Four cycles.
  Interventions: Drug: Irinotecan; Drug: Cisplatin
- Arm B (Active Comparator): Irinotecan 65mg/m2/iv over 90min and cisplatin 30mg/m2/iv over 60min on day 1 and 8, repeat Q 3weeks. Four cycles.
  Interventions: Drug: Irinotecan; Drug: Cisplatin

INTERVENTIONS:
Drug: Irinotecan
Drug: Cisplatin

SUMMARY:
As the gene polymorphism of uridine diphosphate glucuronosyl transferase 1A1(UGT1A1)is related to the side effect of diarrhea induced by irinotecan. UGT1A1 gene *28 (6/6 and 6/7) and *6 (G/G and G/A) is related to low probability of diarrhea and UGT1A1 gene *28 (7/7) and *6 (A/A)is related to high probability of diarrhea. The purpose of this study is to find out the efficacy and side effect between two different dosages of irinotecan combined with cisplatin scheme in extensive disease-small cell lung cancer with UGT1A1 gene *28 (6/6 and 6/7)and *6 (G/G and G/A), based on the hypothesis that the UGT1A1 gene *28 (7/7) and *6 (A/A)is few in the Chinese population and increasing the dose of irinotecan can improve the efficacy without increasing the side effect in the patients with UGT1A1 gene *28 (6/6 and 6/7)*6 (G/G and G/A).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of small-cell lung cancer
* Extensive-stage disease, defined as disease extending beyond one hemithorax involving contralateral mediastinal, hilar or supraclavicular lymph nodes, and/or pleural effusion.
* Males or females between 18 to 75 years
* No prior chemotherapy, if the surgery or radiotherapy has been administered, the interval is at least above four weeks.
* Performance status of 0-2 on the ECOG criteria. Expected survival is above three months.
* At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
* Patient compliance that allow adequate follow-up. Informed consent from patient or patient's relative.
* Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNL x 1.5), and renal (creatinine =< UNL) function
* The gene type of UGT1A1 *28 is 6/6 and 6/7.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.
* No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.

Exclusion Criteria:

* Non small cell lung cancer and carcinoid
* Medically uncontrolled severe diarrhea in recent three weeks.
* Inability to comply with protocol or study procedures.
* Medically uncontrolled serious heart, lung, neurological, psychological, metabolic disease
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Pregnant or breast-feeding.
* Enrollment in other study within 30 days
* Brain metastasis with symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | The first day of treatment to the date that disease progression is reported; assessed up to 3 years

SECONDARY OUTCOMES:
overall survival | the first day of treatment to death or last survival confirm date; assesed up to 3 years
Tumor response rate | Up to 3 years
  the ratio between the number of responders and number of patients assessable for tumor response
Toxicity | the first date of treatment to 30 days after the last dose of study drug
Quality of life | the day before every cycle of chemotherapy; 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Xueqin Yang, M.D., Principal Investigator — Daping Hospital, Third Military Medical University
Locations (3):
- China (3):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Xinan Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality

REFERENCES:
- [Background] Hanna N, Bunn PA Jr, Langer C, Einhorn L, Guthrie T Jr, Beck T, Ansari R, Ellis P, Byrne M, Morrison M, Hariharan S, Wang B, Sandler A. Randomized phase III trial comparing irinotecan/cisplatin with etoposide/cisplatin in patients with previously untreated extensive-stage disease small-cell lung cancer. J Clin Oncol. 2006 May 1;24(13):2038-43. doi: 10.1200/JCO.2005.04.8595. PMID 16648503
- [Background] Gao J, Zhou J, Li Y, Lu M, Jia R, Shen L. UGT1A1 6/28 polymorphisms could predict irinotecan-induced severe neutropenia not diarrhea in Chinese colorectal cancer patients. Med Oncol. 2013;30(3):604. doi: 10.1007/s12032-013-0604-x. Epub 2013 May 18. PMID 23686699
- [Background] Zhang X, Meng X, Wang Y, Yan W, Yang J. Comprehensive analysis of UGT1A1 genetic polymorphisms in Chinese Tibetan and Han populations. Biochem Genet. 2012 Dec;50(11-12):967-77. doi: 10.1007/s10528-012-9536-y. Epub 2012 Sep 16. PMID 22983686
- [Background] Noda K, Nishiwaki Y, Kawahara M, Negoro S, Sugiura T, Yokoyama A, Fukuoka M, Mori K, Watanabe K, Tamura T, Yamamoto S, Saijo N; Japan Clinical Oncology Group. Irinotecan plus cisplatin compared with etoposide plus cisplatin for extensive small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):85-91. doi: 10.1056/NEJMoa003034. PMID 11784874